CLINICAL TRIAL: NCT00093522
Title: A Phase II Pilot Study of Tumor-Loaded Dendritic Cells Alone or Following a Non-Myeloablative Conditioning Regimen in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Vaccine Therapy With or Without Fludarabine in Treating Patients With Stage IV Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Luke's Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000389145; STLMC-IMM-03-05; STLMC-L-03-138
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — FANG vaccine; keyhole-limpet hemocyanin; fludarabine phosphate

INTERVENTIONS:
Biological: autologous tumor cell vaccine
Biological: keyhole limpet hemocyanin
Biological: therapeutic autologous dendritic cells
Drug: fludarabine phosphate
Procedure: conventional surgery

SUMMARY:
RATIONALE: Vaccines made from a person's tumor cells and white blood cells may make the body build an immune response to kill tumor cells. Drugs used in chemotherapy, such as fludarabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining vaccine therapy with fludarabine may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying vaccine therapy and fludarabine to see how well they work compared to vaccine therapy alone in treating patients with stage IV kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the safety of vaccination comprising autologous dendritic cells loaded with autologous tumor lysate and keyhole limpet hemocyanin with vs without non-myeloablative fludarabine in patients with stage IV renal cell carcinoma.
* Compare, preliminarily, the efficacy of these regimens in these patients.
* Compare the overall survival of patients treated with these regimens.

Secondary

* Determine whether this vaccine induces tumor-reactive peripheral T-cell responses or delayed-type hypersensitivity in these patients.

OUTLINE: This is a pilot, randomized study. Patients are randomized to 1 of 2 treatment arms.

All patients undergo surgery to remove tumor at metastatic sites to generate autologous tumor lysate. Patients then undergo leukapheresis to obtain peripheral blood mononuclear cells for the generation of dendritic cells (DC). The DC are then exposed to autologous tumor lysate and keyhole limpet hemocyanin (KLH).

* Arm I: Three weeks after leukapheresis, patients receive vaccination comprising DC loaded with autologous tumor lysate and KLH (DC vaccine) intradermally once every 14 days for a total of 4 injections in the absence of disease progression or unacceptable toxicity.
* Arm II: Two weeks after leukapheresis, patients receive fludarabine IV over 15-30 minutes once daily for 3 days. Beginning approximately 5 weeks after leukapheresis, patients also receive DC vaccine as in arm I.

Patients are followed at 1, 3, and 7-9 weeks, at 4, 6, 9, and 12 months, and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 28 patients (14 per treatment arm) will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Stage IV disease
* Received no benefit from standard therapy OR ineligible for standard therapy OR declined standard therapy
* At least 1 site of metastatic disease that can be surgically removed AND at least 1 site of metastatic disease than can remain in the patient (indicator lesion) after surgery

  * Total volume of the site or sites of disease to be surgically removed must be > 2.0 cm^3
* Unidimensionally measurable disease

  * At least 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No brain metastasis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 6 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 10 g/dL

Hepatic

* SGPT and SGOT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Hepatitis C antibody negative
* Hepatitis B surface antigen negative

Renal

* Creatinine ≤ 1.5 times ULN
* Creatinine clearance > 40 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Immunologic

* Coomb's test negative
* HIV-1 and -2 negative
* No active infection
* No unexplained fever (temperature > 100.5° F or 38.1°C)
* No lymphocytopenia
* No hypogammaglobulinemia
* No autoimmune disease or other immunocompromising condition that would preclude study participation
* No history of impaired immune response
* No history of tuberculosis OR positive PPD skin test
* No history of allergic reaction attributed to compounds of similar biological composition to study vaccine
* No history of allergic reaction to antibiotics

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study participation
* No psychiatric illness or social situation that would preclude study participation
* No other malignancy within the past 5 years except resected basal cell carcinoma or carcinoma in situ of the cervix
* No other concurrent illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* At least 4 weeks since prior steroid therapy or steroid-containing compounds
* At least 2 weeks since prior topical or inhaled steroids

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* See Disease Characteristics

Other

* More than 4 weeks since prior investigational agents
* More than 1 week since prior antibiotics
* No concurrent renal dialysis
* No concurrent anticoagulants
* No other concurrent anticancer agents or therapies
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2004-08

PRIMARY OUTCOMES:
Safety as measured by NCI common toxicity table at completion of study
Response as measured by RECIST guidelines and the Kaplan-Meier method at 5 years
Survival as measured by the Kaplan-Meier method at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John P. Hanson, MD, Principal Investigator — St. Luke's Medical Center
Locations (2):
- United States (2):
  - Midwest Heart Surgery Institute, Limited, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin